CLINICAL TRIAL: NCT04185493
Title: Assessment of Coronary Artery Geometry With Coronary CT Angiography: Evaluation of Atherosclerotic Plaque Burden and Composition
Brief Title: Coronary Artery Geometry and the Severity of Coronary Atherosclerosis
Acronym: GEOMETRY-CTA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Georgios P Rampidis, MD, MSc, Academic Fellow, Aristotle University Of Thessaloniki
Other Study IDs: GEOMETRY_29.01.2019.101068
Record Dates: First submitted 2019-12-01; First posted 2019-12-04 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Coronary Artery Disease; Atherosclerosis; Atherosclerotic Plaque; Stable Angina
Keywords: Geometry; Bifurcation Angle; Cardiac Computed Tomography Angiography; Coronary Artery Disease; Vulnerable Coronary Plaque; Indexed Coronary Volume; Risk Assessment
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis; Plaque, Atherosclerotic; Angina, Stable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CCTA Cohort: Consecutive patients with suspected coronary artery disease and low/intermediate pre-test probability
  Interventions: Diagnostic Test: CCTA

INTERVENTIONS:
Diagnostic Test: CCTA — 128-multislice CT coronary angiography and complex atherosclerotic plaque analysis with the use of CT imaging post-processing techniques.

SUMMARY:
The purpose of this study is to investigate the potential association of coronary artery geometry, based on coronary CT angiography (CCTA), with the complexity and the severity of coronary atherosclerosis.

DETAILED DESCRIPTION:
The angulation of the side branch take-off has been reported to influence the severity of atherosclerosis in coronary bifurcations, as larger angles have been associated with increased plaque burden. Data from computational fluid dynamics studies have confirmed this finding by demonstrating that even in the absence of alterations in the amount of branch flow, a wide angle between the side branches intensifies flow perturbations, increases the spatial endothelial shear stress (ESS) variations in the bifurcation region and the low ESS in the lateral walls, thereby augmenting the atherosclerosis-prone environment. The magnitude of reversed flow, the extension of the recirculation zone and the duration of flow separation during the pulse cycle comprise other haemodynamic parameters which are important in atherogenesis and are amplified by an increased bifurcation angle.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for cardiac CT angiography
* Patients without previous history of Coronary Artery Disease (CAD)
* Age ≥ 18 years
* Patients giving voluntary written consent to participate in the study

Exclusion Criteria:

* Pregnancy or breast-feeding
* Patients with serious concurrent disease and life expectancy of < 1 year
* Patients with a previous history of CAD
* Patients who refuse to give written consent for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients older than 18 years old at entry, of both genders, who referred for coronary CT angiography
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-04 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Left Main Coronary Artery (LMCA) angle of take-off from the aortic root | 30 days
  Measurement using curved Multiplanar Reconstruction (MPR) technique in advantage workstation server
Right Coronary Artery (RCA) angle of take-off from the aortic root | 30 days
  Measurement using curved MPR technique in advantage workstation server
Left Anterior Descending (LAD) / Left Circumflex (LCx) bifurcation angle | 30 days
  Measurement using curved MPR technique in advantage workstation server
Indexed Coronary Volume | 30 days
  Calculated by dividing the total coronary volume to the left ventricle mass, both derived from CCTA (mm3/gr)

SECONDARY OUTCOMES:
Extent of Coronary Atherosclerosis | 30 days
  Total atherosclerotic plaque volume (mm3)
Severity of Coronary Atherosclerosis assessed by using Leiden CTA risk score | 30 days
  Leiden CTA risk score incorporates the presence, extent, severity, location, and composition of coronary artery disease (CAD). Leiden CTA score is calculated using the following approach. First, the presence of CAD is determined in each segment. When plaque is absent the score is 0. When plaque is present a score of 1.1, 1.2 or 1.3 is given according to plaque composition (calcified, noncalcified, and mixed plaque, respectively). Subsequently, this score is multiplied by a weight factor for the location of the segment in the coronary artery tree (0.5 through 6 according to vessel, proximal location and system dominance) and multiplied by a weight factor for stenosis severity (1.4 for ≥50% stenosis and 1.0 for stenosis <50%). The final score (range 0 to 42) is calculated by addition of the individual segment scores.
Severity of Coronary Atherosclerosis assessed by using Gensini score | 30 days
  The relative severity of a lesion is indicated using a score of 1 for 1-25% obstruction and doubling that number as the severity of obstruction progresses with each step in the 25-50-75-90-99-100% diameter reduction. Thus, the severity score for each lesion may range from 1 to 32. Furthermore, the score weighed according to the usual blood flow to the left ventricle in each vessel or vessel segment. A multiplying factor is applied to each lesion score based upon its location in the coronary tree, depending on the functional significance of the area supplied by that segment. If a segment is totally occluded or 99% stenosed and receiving collaterals, a collateral adjustment factor is used, and the adjustment is reduced by the extent of disease in the vessel that is the source of collaterals. The final score is the sum of all the lesion scores.
Complexity of Coronary Artery Disease [CT-SYNTAX score] | 30 days
  CCTA-derived SYNTAX score (CT-SYNTAX score) is a lesion-based grading tool to characterise the coronary vasculature with respect to the number of lesions and their functional impact, location, and complexity. Higher SYNTAX scores, indicative of more complex disease, are hypothesized to represent a bigger therapeutic challenge and to have potentially worse prognosis.
Frequency of occurrence of high-risk plaques | 30 days
  Frequency (%) of occurrence of high-risk plaque features (HU < 30, Remodelling Index > 1.1, napkin-ring sign & spotty calcium)
Plaque burden assessment [Modified Duke CAD Index for coronary CTA] | 30 days
  Patients are assigned a risk score between 0-100 based on former patient prognosis data. The score is an extension of the 3-vessel disease score. It also incorporates stenosis severity and calculates with left main stenosis and proximal left anterior descending stenosis. There is a significant difference between patients' cumulative survival for the different categories. Left main plaque with any additional moderate or severe stenosis indicates the worst outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Haralambos Karvounis, MD, PhD, Study Chair — AHEPA-Department of Cardiology; Konstantinos Kouskouras, MD, PhD, Principal Investigator — AHEPA-Department of Radiology; Georgios Rampidis, MD, MSc, Principal Investigator — AHEPA-Department of Cardiology; Vasileios Rafailidis, MD, PhD, Principal Investigator — AHEPA-Department of Radiology
Locations (1):
- AHEPA University Hospital, Department of Cardiology, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Antoniadis AP, Giannopoulos AA, Wentzel JJ, Joner M, Giannoglou GD, Virmani R, Chatzizisis YS. Impact of local flow haemodynamics on atherosclerosis in coronary artery bifurcations. EuroIntervention. 2015;11 Suppl V:V18-22. doi: 10.4244/EIJV11SVA4. PMID 25983161
- [Background] Rampidis GP, Benetos G, Benz DC, Giannopoulos AA, Buechel RR. A guide for Gensini Score calculation. Atherosclerosis. 2019 Aug;287:181-183. doi: 10.1016/j.atherosclerosis.2019.05.012. Epub 2019 May 10. No abstract available. PMID 31104809
- [Background] Ferencik M. About the twists and turns: Relationship of coronary artery geometry and atherosclerosis. J Cardiovasc Comput Tomogr. 2018 May-Jun;12(3):261-262. doi: 10.1016/j.jcct.2018.04.004. Epub 2018 Apr 24. No abstract available. PMID 29759894
- [Background] Toutouzas K, Benetos G, Karanasos A, Chatzizisis YS, Giannopoulos AA, Tousoulis D. Vulnerable plaque imaging: updates on new pathobiological mechanisms. Eur Heart J. 2015 Dec 1;36(45):3147-54. doi: 10.1093/eurheartj/ehv508. Epub 2015 Sep 28. PMID 26419623
- [Background] Giannopoulos AA, Benz DC, Grani C, Buechel RR. Imaging the event-prone coronary artery plaque. J Nucl Cardiol. 2019 Feb;26(1):141-153. doi: 10.1007/s12350-017-0982-0. Epub 2017 Jul 6. PMID 28685252
- [Background] Kolossvary M, Szilveszter B, Merkely B, Maurovich-Horvat P. Plaque imaging with CT-a comprehensive review on coronary CT angiography based risk assessment. Cardiovasc Diagn Ther. 2017 Oct;7(5):489-506. doi: 10.21037/cdt.2016.11.06. PMID 29255692
- [Background] Pflederer T, Ludwig J, Ropers D, Daniel WG, Achenbach S. Measurement of coronary artery bifurcation angles by multidetector computed tomography. Invest Radiol. 2006 Nov;41(11):793-8. doi: 10.1097/01.rli.0000239318.88270.9f. PMID 17035869
- [Background] Benetos G, Buechel RR, Goncalves M, Benz DC, von Felten E, Rampidis GP, Clerc OF, Messerli M, Giannopoulos AA, Gebhard C, Fuchs TA, Pazhenkottil AP, Kaufmann PA, Grani C. Coronary artery volume index: a novel CCTA-derived predictor for cardiovascular events. Int J Cardiovasc Imaging. 2020 Apr;36(4):713-722. doi: 10.1007/s10554-019-01750-2. Epub 2020 Jan 1. PMID 31894527
- [Background] Benz DC, Benetos G, Rampidis G, von Felten E, Bakula A, Sustar A, Kudura K, Messerli M, Fuchs TA, Gebhard C, Pazhenkottil AP, Kaufmann PA, Buechel RR. Validation of deep-learning image reconstruction for coronary computed tomography angiography: Impact on noise, image quality and diagnostic accuracy. J Cardiovasc Comput Tomogr. 2020 Sep-Oct;14(5):444-451. doi: 10.1016/j.jcct.2020.01.002. Epub 2020 Jan 13. PMID 31974008